CLINICAL TRIAL: NCT00086112
Title: A Double-blind, Randomized, Prospective Study to Evaluate Adjunctive Risperidone Versus Adjunctive Placebo in Generalized Anxiety Disorder Sub-optimally Responsive to Standard Psychotropic Therapy
Brief Title: Study Comparing Risperidone vs Placebo as add-on Therapy in Patients With Generalized Anxiety Disorder Who Are Sub-optimally Responding to Standard Therapy.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Janssen, LP (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR004696
Record Dates: First submitted 2004-06-24; First posted 2004-06-28 (Estimated); Last update posted 2012-07-23 (Estimated); Status verified 2012-07

CONDITIONS: Anxiety Disorders
Keywords: Anxiety; antipsychotic
MeSH Terms: conditions — Anxiety Disorders | interventions — Risperidone

INTERVENTIONS:
Drug: risperidone oral tablets

SUMMARY:
The purpose of this trial is to determine the effectiveness of risperidone as an adjunctive treatment in patients with GAD who demonstrate a less-than-optimal response to their current anxiolytic treatment.

DETAILED DESCRIPTION:
Many patients with Generalized Anxiety Disorder (GAD) do not benefit or show only partial benefit from current psychotropic therapies. This trial was conducted for the purpose of determining the effectiveness of risperidone as an adjunctive treatment in patients with GAD who demonstrate a less-than-optimal response to their current anxiolytic treatment (either allowed antidepressants, benzodiazepines, or buspirone, or combination). Patients were randomized (patients are assigned different treatments based on chance) to either risperidone or placebo for 4 - 6 weeks of double-blind (neither the patient nor the physician knows whether drug or placebo is being taken, or at what dosage) treatment. Patients randomized to risperidone continued on their current anxiolytic treatment (treatment for anxiety) and received risperidone 0.25 mg per day for the first 3 days, 0.5 mg per day for days 4 through 14, and 1 mg per day for days 15 through 28 of the trial. If clinically indicated, on day 29, the dose could be increased to 2 mg per day for the rest of the trial (4 to 6 additional weeks). At each dose level, risperidone was taken by mouth in a single daily dose. Patients were asked questions every one or two weeks, depending on the phase of the trial, to determine efficacy (effectiveness) and safety. The study hypothesis is that risperidone will be more effective as an adjunct to standard psychotropic treatments for symptoms of Generalized Anxiety Disorder than placebo, as measured by a composite of the four most troubling symptoms identified at baseline.

Risperidone 0.25 mg per day for the first 3 days, 0.5 mg per day for days 4 through 14, and 1 mg per day for days 15 through 28 of the trial. If clinically indicated, on day 29, the dose could be increased to 2 mg per day for the rest of the trial (4 to 6 additional weeks). At each dose level, risperidone was taken by mouth in a single daily dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of physical exam
* Treatment with one or more allowed antidepressants and/or anxiety medications for at least the past 8 weeks
* Judgement of the clinician that the patient has shown a sub-optimal response to this treatment
* Current diagnosis of Generalized Anxiety Disorder
* Maintained on a stable, therapeutic dose(s) of the allowed medication(s) for at least the past four weeks

Exclusion Criteria:

* Presence of other serious medical illnesses
* Active use of cocaine or heroin
* History of suicide attempt in past 12 months
* Changes to antidepressant/anti-anxiety regimen (medication or dose) within the four weeks preceding study baseline (Day 1)
* History of clozapine use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in a composite self-rating of the four most troubling symptoms identified at baseline.

SECONDARY OUTCOMES:
Change from baseline and actual values for other efficacy variables (HAM-A, PGIS, CGI-S, SDS, and Q-LES-Q; safety assessment through adverse event reports, laboratory tests, vital signs, physical examinations, and concomitant medications.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Pandina GJ, Canuso CM, Turkoz I, Kujawa M, Mahmoud RA. Adjunctive risperidone in the treatment of generalized anxiety disorder: a double-blind, prospective, placebo-controlled, randomized trial. Psychopharmacol Bull. 2007;40(3):41-57. PMID 18007568
- See also: Study on Adjunctive Risperidone therapy in Generalized Anxiety Disorder That Is Not Responding to Standard Therapy — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=624&filename=CR004696_CSR.pdf